CLINICAL TRIAL: NCT02168595
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Intravenous Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GMI-1271 in Healthy Adult Subjects
Brief Title: Placebo-controlled Single Dose Study to Evaluate Safety and Pharmacokinetics of GMI-1271 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: GMI-1271-101
Record Dates: First submitted 2014-06-17; First posted 2014-06-20 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Healthy Adult Subjects
Keywords: healthy volunteers, GMI-1271
MeSH Terms: interventions — uproleselan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 2 mg/kg GMI-1271 or matching placebo
  Interventions: Drug: GMI-1271; Drug: Placebo
- Cohort 2 (Experimental): 5 mg/kg GMI-1271 or matching placebo
  Interventions: Drug: GMI-1271; Drug: Placebo
- Cohort 3 (Experimental): 10 mg/kg GMI-1271 or matching placebo
  Interventions: Drug: GMI-1271; Drug: Placebo

INTERVENTIONS:
Drug: GMI-1271 — GMI-1271 is a potent, rationally designed glycomimetic E-selectin antagonist
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics of single ascending IV doses of GMI-1271 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending IV dose study conducted at one study center in the United States (US). One (1) cohort of 12 subjects (6 active and 6 placebo) and two (2) cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation. Subjects will participate in only one cohort. Safety will be assessed throughout the study and serial blood samples and urine samples will be collected for the safety and PK assessment of GMI-1271.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or females, 19 to 60 years of age, inclusive.
2. Medically healthy with no clinically significant screening results (e.g., laboratory profiles, medical histories, vital signs, ECGs, physical examination) as deemed by the PI.
3. Females of childbearing potential must either be sexually inactive (abstinent) for 3 months prior to dosing or be using an acceptable birth control method
4. Females must have a negative pregnancy test at the time of screening and prior to dosing for inclusion in the study.
5. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History of any illness that, in the opinion of the PI, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. Hemoglobin level below the lower limit of normal at screening or check-in.
5. Any liver function test (e.g., AST, ALT, bilirubin) 1.5x the upper limit of normal at screening or check-in.
6. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).
7. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
8. Heart rate is lower than 40 bpm or higher than 99 bpm at screening.
9. QTc interval >430 msec for males or >450 msec for females, or history of prolonged QT syndrome.
10. Estimated creatinine clearance < 90 ml/min at screening or check-in.
11. Blood donation or significant blood loss within 56 days prior to dosing.
12. Plasma donation within 7 days prior to dosing.
13. Participation in another clinical trial within 28 days prior to dosing. The 28-day window will be derived from the date of the last study procedure (such as last blood collection or dosing) in the previous study to Day 1 of Period 1 of the current study.

Note: If an increase (>1.5 x N) in bilirubin is present at screening additional liver function tests may be performed (such as ALT, AST, ALP, albumin, and direct and indirect bilirubin) to determine if the increase of bilirubin is due to Gilbert-Meulengracht syndrome. If consistent with Gilbert's syndrome, the Investigator and Sponsor may decide not to consider this as an exclusion. Any such decision will be documented in the study record.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Treatment related adverse events | Day 1-15
  Treatment related adverse events as a measure of safety and tolerability of GMI-1271 (time frame: Day 1-15)

SECONDARY OUTCOMES:
Time of peak plasma concentration (Tmax) | Day 1-3
Pharmacodynamics | Day 1-3
  WBC count, biomarkers to assess pharmacodynamics of single IV dose of GMI-1271 (time frame: Day 1-3)
Peak plasma concentration (Cmax) | Day 1-3
Area under the plasma concentration vs time curve (AUC) | Day 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cook, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Lincoln, Nebraska, United States